



## **INFORMED CONSENT FORM**

## Title

Influence of residual astigmatism on visual acuity in patients undergoing cataract surgery with trifocal intraocular lens implantation

Approved by the CEIm Grupo Hospitalario Quirónsalud-Catalunya on July 29, 2019 (ID: 2019/65-OFT-CMT)



## **STUDY EC042019**

Influence of residual astigmatism on visual quality in patients operated on for cataracts with implantation of trifocal intraocular lenses.

| Me, | (full name of patient) |
|---|---|
| I have read the information sheet give | |
| I have been able to ask questions about | |
| I have received enough information al | |
| I have been informed by the researche | er Enrique Ordiñaga Monreal |
| | s voluntary and that the data will be collected in the |
| conditions detailed in the Patient Info | rmation Sheet. |
| <ul> <li>According to the General Data Prote</li> </ul> | ection Regulation, consent for the processing of your |
| personal data and for its transfer is re- | vocable. You can exercise the right of access, |
| rectification, and cancellation by cont | acting the researcher. |
| <ul> <li>I understand that I can withdraw fro</li> </ul> | m the study: |
| <ul> <li>Whenever you want</li> </ul> | |
| <ul> <li>Without having to explain</li> </ul> | |
| <ul> <li>Without this having an impa</li> </ul> | ct on my medical care |
| <ul> <li>I freely agree to participate in the st</li> </ul> | udy. |
| Patient's Signature | Investigator's Signature |
| Name: | Name: Enrique Ordiñaga |
| Date: | Date: |